CLINICAL TRIAL: NCT02927977
Title: Dry-needling Added to Physical Therapy for Treating Patients With Chronic Non-specific Neck Pain: a Randomized Controlled Trial
Brief Title: Effectiveness of Dry Needling Adding to Physical Therapy in Patients With Chronic Non-Specific Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Fábio Franciscatto Stieven, MsC, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DRY01
Record Dates: First submitted 2016-10-05; First posted 2016-10-07 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Neck Pain
Keywords: dry needling; exercise; manual therapy
MeSH Terms: conditions — Neck Pain; Motor Activity | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Active Comparator): Individuals with neck pain will receive a multimodal rehabilitation program composed by pain education, exercises and manual therapy. Participants will receive 4-6 treatments during 4 weeks.
  Interventions: Other: control
- dry needling (Experimental): Individuals with neck pain will receive a multimodal rehabilitation program composed by pain education, exercises, manual therapy and dry needling in neck muscles. Participants will receive 4-6 treatments during 4 weeks. Participants will receive 4-6 treatments during 4 weeks.
  Interventions: Other: dry needling

INTERVENTIONS:
Other: control — Individuals with neck pain will receive a multimodal rehabilitation program composed by pain education, exercises and manual therapy. Participants will receive 4-6 treatments during 4 weeks.
  Other Names: active control
  Arms: Control
Other: dry needling — Individuals with neck pain will receive a multimodal rehabilitation program composed by pain education, exercises, manual therapy and dry needling in neck muscles. Participants will receive 4-6 treatments during 4 weeks.
  Arms: dry needling

SUMMARY:
The purpose of this randomized clinical trial is to verify the effectiveness of the addition of the dry needling in individuals with non-specific neck pain who receive a multimodal physical therapy rehabilitation program.

DETAILED DESCRIPTION:
Background: Neck pain is a costly and high prevalent problem. Current evidences show that pain education, exercises and manual therapy are recommended to treat patients with chronic non-specific neck pain, but the use of dry needling has not been studied adequately when in combination with these therapies.

Previous trials have shown that dry needling have effectiveness in reducing neck pain in the short and medium term. However, these studies have some limitations as a small sample size and follow-up time reduced. A clinical trial with multimodal treatment method and consistent with clinical practice is needed to determine the effects of dry needling on individuals with non-specific neck pain.

Purpose: The purpose of this randomized clinical trial is to verify the effectiveness of the addition of the dry needling in individuals with non-specific neck pain who receive a multimodal physical therapy rehabilitation program and compare to individuals who received the multimodal physical therapy rehabilitation program without the use of the dry needling.

Design: a randomized single blind placebo controlled trial will be conducted trial in accordance with the CONSORT guidelines. Patients (n=116) with non-specific neck pain will be randomized to receive 1) pain education, manual therapy, and exercise (n=58) or 2) pain education, manual therapy, exercise and dry needling (n=58). Participants will receive 4-6 treatments during 4 weeks. Clinical outcomes (pain intensity, disability,global perceived effect, self-efficacy, quality of sleep and catastrophizing) will be obtained at follow-up appointments at four, twelve and twenty-four weeks after randomisation.

Methods: The primary outcome will be pain (measured by 11-point numerical pain rating scale) and disability (measured by the Neck Disability Index) measure four weeks after randomization. Secondary outcome will be pain and disability in twelve and twenty-four weeks after randomization and global perceived effect (measured by global perceived rating scale), self-efficacy (measured by pain self-efficacy questionnaire), quality of sleep (measure by Pittsburgh quality index), catastrophizing (measure by pain catastrophizing scale) measured four weeks, twelve weeks and twenty-four weeks after randomization and and registration of adverse events (24h, 27h and four weeks after randomization).

Data Analysis: All outcomes will be assessed following intention-to-treat principles. For each outcome, linear mixed models will be employed containing terms for participant, treatment center, group, time and group by time interaction. Known prognostic factors for increased disability in chronic neck pain will be treated as potential confounders and, in the presence of group imbalance despite random allocation, they will be treated as covariates for all outcomes. For the primary outcomes, a p < 0.05 will be considered statistically significant. For all secondary outcomes, a p < 0.01 will be considered statistically significant.

Significance: the results of this study will provide new information about the clinical application of dry needling in additional component for the management of non-specific neck pain.

ELIGIBILITY:
Inclusion Criteria:

* able to speaking and reading in Portuguese, severity of the symptoms at least 3 points on 0-10 numeric pain rating and at least 14% disability on Neck Disability Index.

Exclusion Criteria:

* history of whiplash associated injuries, fibromyalgia, cervical spine symptoms of radiculopathy or myelopathy, use of anticoagulant medication, pregnancy, history of spinal surgeries and "red flags" (spinal fracture, inflammatory diseases, tumor, fracture, rheumatoid arthritis, osteoporosis).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
pain intensity | 4 weeks after randomisation
  measured by 11-point numeric rating scale
disability | 4 weeks after randomisation
  measured by neck disability index

SECONDARY OUTCOMES:
pain intensity | 12, 24 weeks after randomisation
  measured by 11-point numeric rating scale
disability | 12, 24 weeks after randomisation
  measured by neck disability index
global perceived effect | 4,12, 24 weeks after randomisation
  measured by global perceived rating scale
quality of sleep | 4,12, 24 weeks after randomisation
  measure by Pittsburgh quality index
catastrophizing | 4,12, 24 weeks after randomisation
  measure by pain catastrophizing scale
self-efficacy | 4,12, 24 weeks after randomisation
  measured by The Pain Self-Efficacy Questionnaire
adverse events | 24h, 72h and four weeks after randomisation
  record of the adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Fábio F Stieven, Master, Principal Investigator — Federal University of Health Science of Porto Alegre
Locations (1):
- UFCSPA, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided